CLINICAL TRIAL: NCT00006476
Title: A Phase I Study of Intravesicular Suramin in Recurrent Superficial Bladder Cancer
Brief Title: Suramin in Treating Patients With Recurrent Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRC-PHASE I/II-PH1/073; CDR0000068303 (Registry Identifier: PDQ (Physician Data Query)); NCI-954
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-03

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Suramin

INTERVENTIONS:
Drug: suramin
Procedure: conventional surgery

SUMMARY:
RATIONALE: Suramin may stop the growth of bladder cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of suramin in treating patients who have recurrent bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of suramin in patients with recurrent superficial bladder cancer.
* Confirm that there is no significant systemic absorption of this drug when administered intravesically in these patients.

OUTLINE: This is a dose escalation study.

At approximately 14-18 days after surgical resection of bladder tumor(s), patients receive intravesicular suramin via urethral catheter installation into the bladder over 2 hours weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of suramin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients develop dose-limiting toxicity.

Patients are followed at 2-4 weeks.

PROJECTED ACCRUAL: A total of 12-15 patients will be accrued for this study over 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent superficial bladder cancer

  * Intermediate prognosis as defined by the following:

    * Recurrent, multiple Ta, T1 carcinoma
    * Multiple (1-7) tumors
    * Tumors resected previously must be histological grade G1 or G2 OR
* Previously treated superficial bladder cancer requiring followup cystoscopy

  * Recurrent disease diagnosed at surgery
* No tumor invasion into muscle or carcinoma in situ

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm3
* Platelet count at least 150,000/mm3

Hepatic:

* No clinically significant hepatic disease

Renal:

* Creatinine clearance greater than 60 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* No history of adrenal insufficiency
* No other malignancy within the past 5 years except adequately treated cone-biopsied carcinoma in situ of the cervix or nonmelanoma skin cancer
* No history of difficult catheterization
* No confusion or disorientation
* No other condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* No prior radiotherapy to the bladder
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major thoracic or abdominal surgery

Other:

* Recovered from prior therapy and stable for 4 weeks
* At least 6 weeks since prior intravesicular therapy
* No prior or concurrent investigational drugs
* No concurrent anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2000-10; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian L. Harris, MD, Study Chair — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Radcliffe Hospital, Oxford, England, United Kingdom

REFERENCES:
- [Result] Ord JJ, Streeter E, Jones A, Le Monnier K, Cranston D, Crew J, Joel SP, Rogers MA, Banks RE, Roberts IS, Harris AL. Phase I trial of intravesical Suramin in recurrent superficial transitional cell bladder carcinoma. Br J Cancer. 2005 Jun 20;92(12):2140-7. doi: 10.1038/sj.bjc.6602650. PMID 15928663